CLINICAL TRIAL: NCT02206165
Title: A Randomized, Double-blind, Multi-center, Phase 2 Trial to Evaluate the Efficacy and Safety of Candesartan/Amlodipine Combined or Alone and Select Better Dose of CKD-330 in Patients With Essential Hypertension
Brief Title: A Dose Selection Trial of CKD-330 in Patients With Essential Hypertension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 144HT13021
Record Dates: First submitted 2014-06-16; First posted 2014-08-01 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — candesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- Candesartan 8mg + Amlodipine 5mg (Experimental): Candesartan 8mg + Amlodipine 5mg, po, q.d.
  Interventions: Drug: Candesartan 8mg; Drug: Amlodipine 5mg
- Candesartan 8mg + Amlodipine 10mg (Experimental): Candesartan 8mg + Amlodipine 10mg, po, q.d.
  Interventions: Drug: Candesartan 8mg; Drug: Amlodipine 10mg
- Candesartan 16mg + Amlodipine 5mg (Experimental): Candesartan 16mg + Amlodipine 5mg, po, q.d.
  Interventions: Drug: Candesartan 16mg; Drug: Amlodipine 5mg
- Candesartan 16mg + Amlodipine 10mg (Experimental): Candesartan 16mg + Amlodipine 10mg, po, q.d.
  Interventions: Drug: Candesartan 16mg; Drug: Amlodipine 10mg
- Candesartan 8mg (Active Comparator): Candesartan 8mg, po, q.d.
  Interventions: Drug: Candesartan 8mg
- Candesartan 16mg (Active Comparator): Candesartan 16mg, po, q.d.
  Interventions: Drug: Candesartan 16mg
- Amlodipine 5mg (Active Comparator): Amlodipine 5mg, po, q.d.
  Interventions: Drug: Amlodipine 5mg
- Amlodipine 10mg (Active Comparator): Amlodipine 10mg, po, q.d.
  Interventions: Drug: Amlodipine 10mg

INTERVENTIONS:
Drug: Candesartan 8mg — Once a day, 8 weeks
  Arms: Candesartan 8mg; Candesartan 8mg + Amlodipine 10mg; Candesartan 8mg + Amlodipine 5mg
Drug: Candesartan 16mg — Once a day, 8 weeks
  Arms: Candesartan 16mg; Candesartan 16mg + Amlodipine 10mg; Candesartan 16mg + Amlodipine 5mg
Drug: Amlodipine 5mg — Once a day, 8 weeks
  Arms: Amlodipine 5mg; Candesartan 16mg + Amlodipine 5mg; Candesartan 8mg + Amlodipine 5mg
Drug: Amlodipine 10mg — Once a day, 8 weeks
  Arms: Amlodipine 10mg; Candesartan 16mg + Amlodipine 10mg; Candesartan 8mg + Amlodipine 10mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Candesartan/Amlodipine combined or alone and select better dose of CKD-330 in essential hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or above
* Essential hypertension with 90mmHg ≤ mean sitDBP ≤ 115mmHg on target arm at Visit 3
* Ability to provide written informed consent

Exclusion Criteria:

* nean sitDBP ≥ 116mmHg or mean sitSBP ≥ 200mmHg at Visit 1, Visit 2, Visit 3
* The change of mean sitDBP ≥ 10mmHg or mean sitSBP ≥ 20mmHg on target arm at Visit 1
* Known or suspected Stage 2 Hypertension (aortic coarctation, Primary hyperaldosteronism, renal artery stenosis, pheochromocytoma)
* Patients with congestive heart failure(NYHA class III~IV), ischemic heart disease, cardiomyopathy, heart valve disorder, arrhythmia, coronary artery bypass graft
* History of cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months
* Type I Diabets Mellitus, Type II Diabetes Mellitus with HbA1c > 8%
* History of severe or malignant retinopathy
* AST/ALT > UNL * 2, Serum Creatinine > UNL * 1.5, K > 5.5mEq/L
* Patients with acute or chronic inflammatory status, autoimmune disease
* Patients who need to take antihypertensive drug besides Investigational products
* Patients must be treated with medications prohibited for concomitant use during study period
* Hypersensitive to Candesartan/Amlodipine or other dihydropyridine drugs
* Hereditary angioedema or history of angioedema related to ACE inhibitor or angiotensin II receptor blockers
* History of malignant tumor within 5 years
* Patients who are dependent on drugs or alcohol
* History of disability to drug absorption, active inflammatory bowel syndrome with 12months, impaired pancreatic function, GI bleeding, obstructions of urinary tract
* Patients treated with other investigational product within 4 weeks at the time concents are obtained
* Women with pregnant, breast-feeding
* Not eligible to participate for study at the discretion of investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The mean change of sitDBP (sitting diastolic blood pressure) | From baseline at week 8

SECONDARY OUTCOMES:
The mean change of sitDBP | From baseline at week 4 and week 8
The mean change of sitSBP | From baseline at week 4 and 8
Responder rate: The change of sitDBP > 10mmHg, sitSBP > 20mmHg | From baseline at week 4 and 8
Control rate: Patient achieving sitDBP < 90mmHg and sitSBP < 140mmHg | At week 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Cheol-Ho Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea